CLINICAL TRIAL: NCT01878240
Title: Prevention of Type II Endoleaks During Endovascular Treatment of Abdominal Aortic Aneurysm: Endovascular Treatment Versus Combination With Coil Embolisation of the Aneurysmal Sac
Acronym: SCOPE1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Collaborators: Institut Mutualiste Montsouris (Other); Henri Mondor University Hospital (Other); Unité de Recherche Clinique du Centre chirurgical marie Lannelongue (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P12-37813003/2012A01258-35; IDRCB 2012-A0125-35 (Other: P12-37813003)
Record Dates: First submitted 2013-05-17; First posted 2013-06-14 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2019-04

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Vascular surgery; Abdominal Aortic aneurysm; endovascular
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EVAR (Active Comparator): Endovascular repair of an Abdominal Aortic Aneurysm
  Interventions: Procedure: EVAR without coils embolization/ Coils embolization during EVAR
- Coil embolization during EVAR (Experimental): coil embolization during Endovascular repair
  Interventions: Procedure: EVAR without coils embolization/ Coils embolization during EVAR

INTERVENTIONS:
Procedure: EVAR without coils embolization/ Coils embolization during EVAR
  Other Names: Coil embolization during endovascular Aortic Abdominal Aneurysm repair

SUMMARY:
Abdominal aortic aneurysms (AAAs) continue to be a leading cause of death in older age groups. In the 60-85 year-old population, AAA represents the 14th-leading cause of death. Federal funding through Medicare has been allocated for early detection using abdominal ultrasound screening programs. Despite these more aggressive screening programs and concerted efforts by surgeons for timely repair, the incidence of ruptured AAA has continued to increase.

Endovascular aneurysm repair (EVAR) has been the most common type of repair since 2006. Multiple studies reflecting decreased perioperative morbidity and mortality over open repair make this an attractive option for patients. EVAR requires more intensive follow-up than standard open surgical repair, however. Secondary interventions are more common to maintain "seal" of the endograft within the aorta and subsequent exclusion of the aneurysmal component.

The term endoleak is specific to EVAR, and describes the primary means by which endografts fail. Type I endoleaks occur because of inadequate graft seal proximally or distally, resulting in perigraft flow and aneurysm sac pressurization. Type II endoleaks occur when branch arteries arising from the aneurysmal aorta back-bleed into the aneurysm sac due to collateral flow. Type III endoleaks occur when flow persists between segments of a modular graft. Type IV endoleaks occur when flow persists through endograft material (graft porosity). Type V endoleaks have also been called "endotension", and occur when pressurization of the sac occurs in the absence of any demonstrable endoleak. Type I and Type III endoleaks are most concerning for rupture, although persistent Type II endoleaks can also lead to aneurysm rupture and premature death.

The most common method of EVAR follow-up is computed tomographic angiography (CTA). These studies allow accurate measurement of aneurysm sac diameters and volumes. They also are highly sensitive and specific for endoleaks. Type II endoleaks are treated if they remain persistent and are present in the setting of aneurysm sac enlargement. Type I and III endoleaks are immediately treated when identified. Type IV endoleaks are rarely seen with current endograft technology.

DETAILED DESCRIPTION:
Study Objectives:

The purpose of the current study is to compare the level of endoleaks between group 1 and 2 at 1, 6, 12 and 24 months.

Study Design Prospective interventional study, multicenter, open, randomized trial comparing the type II endoleak level in patients who benefited the endovascular AAA repair (group 1: without coils) versus combination with coil embolization of the aneurysmal sac (group II: with coils).

The choice of treatment is randomized.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Carrying a sub-renal AAA with a diameter of at least 5 cm at a rate of growth or greater 1cm/an diameter (according to Haute Autorité de Santé (HAS) recommendations toE VAR treatment),
* Patients with high risk of type II endoleak (clouding of an aortic aneurysm sac by collateral branch), respondents with at least one of the following criteria on the scanner to be included:

  * The presence of a pair of permeable lumbar arteries.
  * The presence of a patent inferior mesenteric artery.

Exclusion Criteria:

* Sub renal Collet <10 mm
* Angulated > 60 °
* No collateral arising from the aneurysmal sac
* Iliac aneurysms associated
* Ruptured AAA
* Pregnant Women
* Lack of consent
* Lack of social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-05 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Evaluation at one month the presence or absence of endoleak type II in all patients for each group by Computer Tomography and Doppler. | 1 month

SECONDARY OUTCOMES:
• Evaluation at 6, 12 and 24 months by CT and doppler: -The rate of type II endoleak | 6, 12 and 24 months
• Mortality and morbidity . | 1, 6, 12 and 24 months
• Number of additional procedures -endovascular -surgical | 1, 6, 12 and 24 months
• Complications of endovascular procedures away from the EVAR -Thrombosis of leg -Limb occlusion -Evolution of the aneurysmal neck | 1, 6, 12 and 24 months
• Monitoring of renal function (creatinine clearance). | 1, 6, 12 and 24 months
• Evaluation at 6, 12 and 24 months by CT and doppler: -Measurement of the maximum transverse aneurysm diameter | 6, 12 and 24 months
• Evaluation at 6, 12 and 24 months by CT and doppler: -volumetric measurement of the sac aneurysmal | 6, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Dominique FABRE, Vascular surgeon, Principal Investigator — Centre Chirurgical Marie Lannelongue
Locations (3):
- France (3):
  - Hopital Henri Mondor - APHP, Créteil, Île-de-France Region
  - Centre Chirurgical MarieLannelongue, Le Plessis-Robinson, Île-de-France Region
  - Institut Mutualiste Montsouris, Paris, Île-de-France Region

REFERENCES:
- [Result] Lederle FA, Freischlag JA, Kyriakides TC, Matsumura JS, Padberg FT Jr, Kohler TR, Kougias P, Jean-Claude JM, Cikrit DF, Swanson KM; OVER Veterans Affairs Cooperative Study Group. Long-term comparison of endovascular and open repair of abdominal aortic aneurysm. N Engl J Med. 2012 Nov 22;367(21):1988-97. doi: 10.1056/NEJMoa1207481. PMID 23171095
- [Result] Jackson RS, Chang DC, Freischlag JA. Comparison of long-term survival after open vs endovascular repair of intact abdominal aortic aneurysm among Medicare beneficiaries. JAMA. 2012 Apr 18;307(15):1621-8. doi: 10.1001/jama.2012.453. PMID 22511690
- [Result] Stather PW, Sidloff D, Dattani N, Choke E, Bown MJ, Sayers RD. Systematic review and meta-analysis of the early and late outcomes of open and endovascular repair of abdominal aortic aneurysm. Br J Surg. 2013 Jun;100(7):863-72. doi: 10.1002/bjs.9101. Epub 2013 Mar 8. PMID 23475697
- [Result] Piazza M, Frigatti P, Scrivere P, Bonvini S, Noventa F, Ricotta JJ 2nd, Grego F, Antonello M. Role of aneurysm sac embolization during endovascular aneurysm repair in the prevention of type II endoleak-related complications. J Vasc Surg. 2013 Apr;57(4):934-41. doi: 10.1016/j.jvs.2012.10.078. Epub 2013 Feb 4. PMID 23384494
- [Result] Schanzer A, Greenberg RK, Hevelone N, Robinson WP, Eslami MH, Goldberg RJ, Messina L. Predictors of abdominal aortic aneurysm sac enlargement after endovascular repair. Circulation. 2011 Jun 21;123(24):2848-55. doi: 10.1161/CIRCULATIONAHA.110.014902. Epub 2011 Apr 10. PMID 21478500
- [Derived] Fabre D, Mougin J, Mitilian D, Cochennec F, Garcia Alonso C, Becquemin JP, Desgranges P, Allaire E, Hamdi S, Brenot P, Bourkaib R, Haulon S. Prospective, Randomised Two Centre Trial of Endovascular Repair of Abdominal Aortic Aneurysm With or Without Sac Embolisation. Eur J Vasc Endovasc Surg. 2021 Feb;61(2):201-209. doi: 10.1016/j.ejvs.2020.11.028. Epub 2020 Dec 17. PMID 33342658